CLINICAL TRIAL: NCT00273507
Title: Neoadjuvant Chemotherapy in Resectable NSCLC Stages IB, IIA, IIB, and IIIA/T3 But Not IIIA/N2
Brief Title: Neoadjuvant Chemotherapy in Non Small Cell Lung Cancer (NSCLC) Stages IB, IIA, IIB, and IIIA/T3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neoadjuvant treatment in NSCLC
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; neoadjuvant; resection
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel

INTERVENTIONS:
Drug: Carboplatin and Paclitaxel

SUMMARY:
Randomised trial of chemotherapy or not before surgery in early resectable stages of NSCLC (IB, IIA, IIB, and IIIA/N2).

DETAILED DESCRIPTION:
Randomisation between 3 courses of neoadjuvant Carboplatin plus Paclitaxel or no chemotherapy before surgery.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC
* Stages IB, IIA, IIB, IIIA/T3
* Lung function test allowing surgery
* Age 18-75 years

Exclusion Criteria:

* Poor lung function
* Performance status 3-4
* Mediastinal lymph node involvement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 1998-01; Study Completion 2006-01

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
Time to progression
Complete resection rate

CONTACTS AND LOCATIONS:
Overall Officials: Jens B. Sorensen, MD, Study Chair — Dept. Oncology, Rigshospitalet
Locations (1):
- Dept. Oncology, Rigshospitalet, Copenhagen, Copenhagen, Denmark